CLINICAL TRIAL: NCT03348033
Title: Adoptive Immunotherapy in Patients With Chronic Myeloid Leukemia: Phase I/II Study to Test the Safety and Feasibility of Autologous Activated and Expanded Natural Killer Cells
Brief Title: Safety and Feasibility of the Use of Natural Killer Cells in Patients With Chronic Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160409
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic Myeloid Leukemia + NK cell (Experimental): Starting on Day -7, G-CSF daily by vein until post nadir of absolute neutrophil counts (ANC) are equal or over 1000. Day -6 to Day -2 Fludarabine administrated by vein at 30 mg/m^2. Four hours later Cytarabine administrated by vein at 2 g/m^2. Natural killer (NK) cell infusion Days 0 to 14 for 6 doses total.
  NK Cell infusion on Days 0 to 14 for 6 doses total.
  Interventions: Biological: Chronic Myeloid Leukemia + NK cell

INTERVENTIONS:
Biological: Chronic Myeloid Leukemia + NK cell — Patients with chronic phase chronic myeloid leukemia who lost response to the second line of treatment with tyrosine kinase inhibitor with indication of bone marrow transplantation or refractory. Infusion of autologous natural killer cells, expanded in the laboratory, after chemotherapeutic conditioning.

SUMMARY:
The purpose of this study is to evaluate safety, feasibility and maximum tolerated dose of NK cells cultured in vitro as adjuvant treatment of patients with chronic myeloid leukemia candidates to allogenic bone marrow transplantation or refractory to conventional treatment.

DETAILED DESCRIPTION:
Natural killer (NK) cells are one of the main type of immune cells that mediate the graft-versus-leukemia (GVL) effect. They are a fundamental part of innate immunity, with a major role in rapid response against infectious agents and activating immune system against tumoral cells. Patients with chronic myelogenous leukemia (CML), however, seem to have lower NK cell counts as disease progresses from chronic phase to blast crisis, as well as diminished cytotoxicity in those NK cells remaining. Therapeutic role of the NK cell ability to target certain specific cells is currently being studied, especially regarding their action against tumoral cells. Chronic myeloid leukemia studies with NK cells have so far demonstrated that autologous ex vivo activated NK cells are able to suppress in vitro the presence of the breakpoint cluster region-abelson leukemia virus (BCR-ABL) oncogene. These studies have demonstrated that adoptive NK cell therapy may have a potential role in treatment of CML patients.

The purpose of this study is to evaluate safety, feasibility and maximum tolerated dose of NK cells cultured in vitro as adjuvant treatment of patients with chronic myeloid leukemia candidates to allogenic bone marrow transplantation or refractory to conventional treatment.

NK cells will be expanded from peripheral blood mononuclear cells after depletion of T cells. They ar going to be co-cultured with clone 9 K562 artificial antigen presenting cell (aAPCs), which are posteriorly modified to also express membrane interleukin-21 (mIL-21)

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic phase CML who lost response to the second line of treatment with tyrosine-kinase inhibitor (TKI) with indication for bone marrow transplantation.
* Accelerated phase patients who are candidates for bone marrow transplantation.
* Patient with CML in blast crisis.
* Patient aged between 2 and 59 years.
* patient should have recovered from the toxicity related to previous treatment of cytotoxic agents received within 4 weeks before starting treatment in this protocol, except for cytopenias resulting from persistent disease and alopecia, or non-haematological toxicities grades 1 and 2

Exclusion Criteria:

* Zubrod performance scale ≥ 2
* Renal impairment: Serum creatinine> 2mg / dL for adults and> 2mg / dL or> 2 times the upper limit of normality for age (whichever is less) for children.
* Impaired hepatic function, defined as: total bilirubin> 2 mg / dL and alanine aminotransferase (ALT) 2.5 times upper limit of normal for age (unless Gilbert's disease or abnormal liver function due to primary disease).
* Pulmonary symptoms with pulse oximetry <92%.
* Congestive Heart Failure Classification New York Heart Association> III
* Positive serological test for pregnancy within two weeks prior to enrollment in women of childbearing potential (non-fertile age defined as pre-menarche, post-menopausal over one year, or surgically sterilized).
* Positive serology for human immunodeficiency virus (HIV).
* Have undergone investigational therapies in four weeks prior to treatment begin under this protocol.
* Congestive heart failure < 6 months prior to screening.
* Unstable angina < 6 months before screening.
* Myocardial infarction < 6 months prior to selection.
* Non-signing of the informed consent.

Ages: 2 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of membrane-bound interleukin 21 (mbIL21)-Expanded Haploidentical NK Cells After Induction Chemotherapy with Fludarabine, Cytarabine, and Granulocyte-colony stimulating factor (G-CSF) | 28 days
  Maximum tolerated dose defined as highest dose studied in which 6 patients have been treated and at most 2 patients with dose-limiting toxicities (DLTs) observed.
  A dose-limiting toxicity (DLT) is defined as:
  Acute severe (grade 3 or 4) infusional allergic reaction related to the NK cells infusion.
  Prolonged cytopenia beyond D+28. If neutropenia is still present at day 28, that will trigger the designation of prolonged neutropenia as a DLT. If neutrophil counts have recovered by day 28, then no DLT will have occurred. In either case, the status of neutrophil recovery beyond day 28 will not change the designation of DLT or No DLT made at day 28.
  Acute graft-versus-host disease (GvHD) overall grade 3 or 4. Severe (grade 3 or 4) unexpected toxicity related to the NK cell infusion

SECONDARY OUTCOMES:
Molecular response Assessment Following Infusion of the NK Cells | Baseline up to Day 56
  Percentage of participants with major molecular response - amount of BCR-ABL gene in the blood is 1/1000th (or less) of what is expected in someone with untreated CML.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Silla, Physician, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Centro Terapia e Tecnologia Celular, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided